CLINICAL TRIAL: NCT03442335
Title: Implantation Test for Endometrial Receptivity
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: RG_17-179; 233994 (Other: IRAS)
Record Dates: First submitted 2018-01-30; First posted 2018-02-22 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2020-11

CONDITIONS: Pregnancy Loss; Miscarriage
Keywords: embryo implantation; endometrial receptivity; chromohysteroscopy; transcriptomics; proteomics; metabolomics; implantation window; luteal phase
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endometrial samples taken during the implantation window (mid luteal phase, timed based on LH surge).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recurrent miscarriage: 2+ miscarriages: Women who suffered 2 or more unexplained recurrent miscarriages.
  Interventions: Diagnostic Test: Chromohysteroscopy; Diagnostic Test: Endometrial biopsy (Pipelle)
- Extreme recurrent miscarriage: 5+ miscarriages: Women who suffered 5 or more unexplained recurrent miscarriages.
  Interventions: Diagnostic Test: Chromohysteroscopy; Diagnostic Test: Endometrial biopsy (Pipelle)

INTERVENTIONS:
Diagnostic Test: Chromohysteroscopy — Standard hysteroscopy followed by injection of a dye, in this case iodine.
Diagnostic Test: Endometrial biopsy (Pipelle) — A narrow plastic tube (Pipelle) is passed through the cervix to aspirate a sample of endometrial tissue.
  Other Names: Endometrial sampling

SUMMARY:
Background Miscarriage is the most frequent complication of pregnancy and represents the spontaneous loss of the embryo or foetus before it is able to survive independently (24 weeks of gestation). It affects up to 50% of pregnancies with the vast majority (80%) occurring at pre-clinical stage before the woman recognises the pregnancy. Up to 5% of couples suffer recurrent miscarriage defined as 2-3 or more miscarriages leading to physical, emotional and financial consequences for couples, doctors and medical systems.

Different maternal health problems (thyroid disease, sticky blood, autoimmune disease, anatomical anomalies of the womb) and embryo defects may be responsible for some of the miscarriages; however, more than 50% of the occurrences have no identifiable cause based on the current diagnostic tests.

Aim The aim of the present research proposal is to understand the role of the lining of the womb in miscarriage and to explore the development of a potential implantation test that is cost-effective and may be implemented in clinical practice.

Methods Over a period of two years, women who suffered recurrent miscarriage will be approached in the advanced miscarriage clinic at Birmingham Women's Hospital during their routine appointment. Participants will be invited to participate by undergoing chromohysteroscopy and/or a biopsy from the lining of the womb during an outpatient appointment.

Chromohysteroscopy is based on a routine hysteroscopy which involves visualising the inside of the womb using a narrow telescope passed through the neck of the womb (cervix). "Chromo" comes from the fact that an iodine based dye will be injected to increase the power of the test.

The biopsy will be taken using a narrow plastic tube passed through the cervix. It is a standard diagnostic test for women with abnormal bleeding. As part of the present research, different cells and molecules will be analysed from the biopsy sample.

DETAILED DESCRIPTION:
The Tommy's National Centre for Miscarriage Research in Birmingham is a Research Centre which brings together an interdisciplinary translational medicine research grouping jointly at the Birmingham Women's and Children's NHS Foundation Trust (BWCNFT) and the University of Birmingham (UoB). The overarching Tommy's Centre funding includes sites at the University of Warwick and Imperial College London. The Centre is dedicated to research across all aspects of miscarriage and early pregnancy complications including basic scientific, medical, social and ethical issues.

This research project will occur alongside an advanced miscarriage clinic at Birmingham Women's Hospital. The Study Office belongs to the University of Birmingham and is located within the Birmingham Women's Hospital (Academic Department, 3rd floor). Computers are linked to the University's Network and all the electronic data will be held within this network.

The research project is divided into a number of three work packages and the findings from these will build on each other. Therefore, we have incorporated each of these distinct work packages within this research project protocol, with methodological details and objectives of each.

Work package 1: Target Product Profile (TPP) The TPP will convey information regarding the proposed use, context of use, patients' and clinicians' needs for an endometrial test in relation to endometrial receptivity, recurrent miscarriage and recurrent implantation failure.

Women who suffer recurrent miscarriage are referred for routine care to the Recurrent Miscarriage Clinic within Birmingham Women's Hospital by their GP or by other NHS Early Pregnancy Units. Women attending the Recurrent Miscarriage Clinic will be invited to fill in a questionnaire during their waiting time prior to the consultation by one of the research nurses who work within the Recurrent Miscarriage Clinic. The purpose of the questionnaire is to gain insight into women's view and expectations in relation to a new endometrial receptivity test.

Work package 2: Chromohysteroscopy Hysteroscopy is the procedure in which the uterine cavity is viewed using a hysteroscope (lighted scope) inserted through the cervix. It is used routinely in the NHS for women with varying indications (ie: polyps or fibroids suspected on ultrasound, thin endometrium, adhesions etc). In addition to morphologic abnormalities (ie: septum, polyps, adhesions), hysteroscopy may identify direct visual appearances relevant to endometrial receptivity.

Chromohysteroscopy involves flushing the endometrial surface with a dye (ie: methylene blue) in order to increase the sensitivity of hysteroscopy for the diagnosis of subtle endometrial pathologies which have not produced macroscopic changes.

All previous chromohysteroscopic studies used methylene blue as a dye to enhance the visibility of endometrial abnormalities based on the ability of necrotic endometrial cells to absorb/retain the dye. The investigators plan to further develop this approach by using iodine in relation to the known endometrial properties.

It is well known that iodine interacts with glycogen to generate a brown-blue colour. The glycogen-iodine reaction normally enables the identification of high vaginal and cervical lesions during colposcopic examinations that women undergo routinely in the NHS when there is a suspicion on their smear tests.

The investigators hypothesise that aberrations in the secretory phase of the endometrial development may be identified using iodine chromohysteroscopy based on the interaction between iodine and glycogen which generates a brown-blue colour.

Work package 3: OMICS studies on endometrial samples Omics- refer to the application of high-throughput techniques which simultaneously examine changes in different molecular compartments: genomics, transcriptomics, proteomics, metabolomics etc. The understanding of human endometrial physiology and pathophysiology is being revolutionised by the use of omics-; however, current understanding of different complex phenotypes related to fertility remains incomplete, inconsistent and without strong clinical application.

A Pipelle biopsy of the endometrium involves passing a narrow plastic tube through the cervix to obtain a sample by aspiration. It is routinely used in the NHS to rule out endometrial hyperplasia/carcinoma in women suffering from heavy menstrual bleeding or postmenopausal bleeding.

The investigators hypothesise that women who suffered recurrent reproductive failure may have altered transcriptomics, proteomics, and metabolomics profiles in their endometrium. Identifying these changes may provide diagnostic and prognostic markers for future pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with unexplained recurrent miscarriage (2+ miscarriages with negative standard miscarriage investigations)
* regular menstrual cycles

Exclusion Criteria:

* women who have irregular menstrual cycles or those who require fertility treatments
* any positive finding or health issue that may explain the diagnosis of recurrent miscarriage
* women who are pregnant at the time of the study investigations
* women who are participants in other interventional studies or trials

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women who suffered recurrent miscarriage (2+ miscarriages).
Study Population: A cohort of women who suffered unexplained recurrent miscarriage will be sub grouped in two study populations: women who suffered two or more miscarriages and women who suffered five or more miscarriages (extreme recurrent miscarriage cohort). A total of 60 women will be recruited for the study investigations (30 for chromohysteroscopy and 30 for endometrial biopsy).
  We will select a very narrow phenotype in order to increase the study's sensitivity and power. Participants will be 18-35 years old, not pregnant and regularly menstruating in order to reduce the age effect on the pregnancy outcome. They will be diagnosed as having unexplained recurrent miscarriage by undertaking the standard miscarriage investigations.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Iodine absorption | 2 years
  Iodine interaction with the mid luteal phase endometrium.
Transcriptome profile | 2 years
  Transcriptomics analysis of endometrial samples.
Proteome profile | 2 years
  Proteomics analysis of endometrial samples.
Metabolome profile | 2 years
  Metabolomics analysis of endometrial samples.

SECONDARY OUTCOMES:
Miscarriage rate | 5 years
  Miscarriage rates in future pregnancies.
Live birth rate | 5 years
  Live birth rates in future pregnancies.

CONTACTS AND LOCATIONS:
Overall Officials: Laurentiu Craciunas, Study Chair — Tommy's National Centre for Miscarriage Research
Locations (6):
- United Kingdom (6):
  - Tommy's National Centre for Miscarriage Research, Birmingham
  - North Bristol NHS Trust, Bristol
  - Countess of Chester Hospital HNS Foundation Trust, Chester
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Saint Mary's Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request by December 2027.

REFERENCES:
- [Result] Craciunas L, Pickering O, Chu J, Zurauskiene J, Coomarasamy A. Target Product Profile for an endometrial receptivity test: women's perspective. Eur J Obstet Gynecol Reprod Biol. 2020 Oct;253:42-47. doi: 10.1016/j.ejogrb.2020.07.058. Epub 2020 Aug 1. PMID 32771887
- [Result] Craciunas L, Pickering O, Chu J, Choudhary M, Zurauskiene J, Coomarasamy A. The transcriptomic profile of endometrial receptivity in recurrent miscarriage. Eur J Obstet Gynecol Reprod Biol. 2021 Jun;261:211-216. doi: 10.1016/j.ejogrb.2021.04.041. Epub 2021 Apr 30. PMID 33971384
- [Result] Craciunas L, Chu J, Pickering O, Mohiyiddeen L, Coomarasamy A. The metabolomic profile of endometrial receptivity in recurrent miscarriage. Minerva Obstet Gynecol. 2023 Dec;75(6):526-534. doi: 10.23736/S2724-606X.22.05151-X. Epub 2022 Oct 4. PMID 36193833